CLINICAL TRIAL: NCT04557813
Title: Registry for Molecular Testing, Treatment and Outcome of Patients With Locally Advanced or Metastatic Solid Tumors Harboring a Fusion of NTRK1, NTRK2 or NTRK3
Brief Title: Registry for Molecular Testing, Treatment and Outcome of Patients With Solid Tumors Harboring a NTRK Gene Fusion
Acronym: REALTRK
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-040444
Record Dates: First submitted 2020-09-02; First posted 2020-09-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: NTRK Family Gene Mutation
Keywords: NTRK; NTRK-fusion; Neurotrophic Tyrosine Receptor Kinase; NTRK Gene Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IC before start of any treatment: Informed consent (IC) before start of any treatment after diagnosis of NTRK fusion-positive cancer. All data after diagnosis of NTRK fusion-positive cancer are collected prospectively.
- IC after start of any treatment: IC after start of any treatment after diagnosis of NTRK fusion-positive cancer. Data after study inclusion are collected prospectively and retrospectively.
- Deceased patients: Patients deceased prior to study inclusion (no IC required). All data are collected retrospectively.

SUMMARY:
The objective of this registry is to analyze treatment reality and outcome of patients with locally advanced or metastatic solid tumors harboring a fusion of NTRK1, NTRK2 or NTRK3

DETAILED DESCRIPTION:
The REALTRK registry will provide data on treatment reality of patients with locally advanced or metastatic solid tumors harboring NTRK1, NTRK2 or NTRK3 gene fusions, thereby generating real world evidence. It will identify factors that influence treatment decisions after receiving the diagnosis of a NTRK (Neurotrophic Tyrosine Receptor Kinase) fusion-positive cancer. All treatment lines administered before and after the molecular diagnosis of a NTRK fusion-positive cancer, irrespective of the type of antineoplastic treatment, will be documented. Data will be assessed at least 36 months per patient (i.e. until 36 months after inclusion of the last patient in the study). This approach will allow a description of TRK fusion protein-targeted therapies and other therapy strategies regarding effectiveness and disease-related symptomology within the limitations of non-randomized studies in terms of comparative analyses. Intra-individual and inter-individual comparisons (for the latter, provided that a sufficient number of patients with a NTRK fusion-positive cancer are not treated with a TRK inhibitor) could be performed.

The associated biomarker profiling module of the REALTRK registry will aim to set up a decentralized biobank for future research on molecular alterations.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic solid tumor with a documented NTRK gene fusion, based on a validated assay (according to current ESMO recommendations), or the provision of tumor material for central retesting
* Molecular pathology or molecular diagnostics report with details on NTRK gene fusion testing must be available
* Aged ≥ 18 years
* Signed and dated informed consent form (ICF) (only if patient is alive at time of data entry into the project; not applicable for inclusion of deceased patients' data)

Exclusion Criteria:

* Treatment with a TRK inhibitor prior to Sept 19th, 2019 (Germany) or May 28th, 2020 (Switzerland)
* Participation in a clinical trial with a TRK inhibitor before or at enrolment (liv-ing patients) or before inclusion (deceased patients)
* Deceased patients who have explicitly contradicted further use of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced (locally advanced or metastatic) solid tumors harboring a NTRK1, NTRK2 or NTRK3 gene fusion
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response rate | through study completion, at least 1 year
  Proportion of patients with CR or PR as best response

SECONDARY OUTCOMES:
Patient and disease characteristics | through study completion, at least 1 year
  Descriptive summary of demographics, patient and disease characteristics
Test methods used for diagnosis of a NTRK fusion-positive cancer | Day 1
  Description of test methods used for diagnosis of a NTRK fusion-positive cancer and results thereof
Physician-reported factors affecting decision to test for NTRK fusion and treatment decision | Day 1
  Description of physician-reported factors affecting decision to test for NTRK fusion and treatment decision making after diagnosis of NTRK gene fusion
Treatment reality after diagnosis of NTRK gene fusion | through study completion, at least 1 year
  Description of all treatment lines given to the patient after diagnosis of NTRK gene fusion including: Type of treatment (Systemic TRK inhibitor treatments or Non-TRK inhibitor treatments), treatment duration, dosing, treatment modifications and reasons thereof, reasons for end of treatment.
Safety of TRK inhibitor treatments | through study completion, at least 1 year
  Treatment-emergent AEs (i.e., AEs which occurred during a specific TRK inhibitor treatment and in the respective survival FU) will be calculated per patient (absolute and relative frequencies) and case-based (absolute frequencies). The occurrence of any (S)AE will be displayed overall and per CTCAE grade. Adverse drug reactions (ADRs) and AESIs will be displayed accordingly.
  Incidence of AEs (MedDRA Preferred Term (PT) by System Organ Class (SOC)) will be calculated accordingly for each type of AE/ADR.
Physician-reported evaluation of TRK inhibitor therapy | Day 1
  Description of physician-reported evaluation of TRK inhibitor therapy
Disease-related symptoms | through study completion, at least 1 year
  Description of courses of disease-related symptoms (weight loss, ECOG) after diagnosis of NTRK gene fusion (Only for patients of inclusion group I)
Disease control rate | through study completion, at least 1 year
  Proportion of patients with CR, PR or SD as best response
Time to Response | through study completion, at least 1 year
  Time from start of treatment to the first objective tumor response (e.g., tumor shrinkage of ≥30%) observed for patients who achieved a CR or PR
Duration of Response | through study completion, at least 1 year
  Time from documentation of tumor response to disease progression or death from any cause
Progression-free survival | through study completion, at least 1 year
  Time from start of treatment until disease progression or death
Overall Survival | through study completion, at least average of 1 year
  Time from start of treatment until death of any cause
PFS ratio | through study completion, at least 1 year
  ratio of PFS of the first treatment line with a TRK inhibitor to time to progression (TTP) in the preceding treatment line without a TRK inhibitor
Event-free survival | through study completion, at least 1 year
  Time from start of treatment until PD or death

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kasenda, PD Dr. Dr., Study Director — Universitätsspital Basel, Petersgraben 4, 4031 Basel, Switzerland
Locations (26):
- Germany (25):
  - Universitätsklinikum Augsburg, Augsburg
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Gesundheit Nord, Klinikverbund Bremen, Bremen
  - PIOH - Praxis Internistische Onkologie und Hämatologie, Cologne
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Asklepios Klinik Altona, Hamburg
  - Onkologische Schwerpunktpraxis, Hanover
  - Gemeinschaftspraxis, Hanover
  - SLK Kliniken Heilbronn Klinik für Innere Medizin III, Heilbronn
  - Klinikum Kempten, Kempten
  - Asklepios MVZ Bayern, Schwerpunkt Hämatologie/Onkologie, Landsberg
  - Onkologische Praxis am Marien-Krankenhaus, Lübeck
  - Praxis für Onkologie, Mönchengladbach
  - Klinikum rechts der Isar der TUM Innere Medizin II, München
  - Universitätsklinikum Münster, Medizinische Klinik A, Münster
  - TZN - Tumorzentrum Niederrhein GmbH, Neuss
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Praxis und Tagesklinik für Onkologie und Hämatologie, Recklinghausen
  - Klinikum Rosenheim, Rosenheim
  - Zentrum Ambulante Onkologie, Schorndorf
  - MVZ Kloster Paradiese GbR, Soest
  - MVZ für Hämatologie und Onkologie, Ulm
  - Onkologie Schwarzwald-Alb, Villingen-Schwenningen
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No